CLINICAL TRIAL: NCT02860637
Title: Level and Degree of Spinal Cord Injury and Its Impact on Male Sexual Function
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Josepha Karinne de Oliveira Ferro, Psysical Therapist, Universidade Federal de Pernambuco
Other Study IDs: Spinal Cord and sexuality
Record Dates: First submitted 2016-07-31; First posted 2016-08-09 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Spinal Cord Injury
Keywords: Sexuality; Spinal cord injuries; Penile erection; erectile dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality; Erectile Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionnaires — Sexual function was assessed by the International Index of Erectile Function (IIEF) and level and degree of injury were determined following the guidelines of the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury.

SUMMARY:
In addition to the motor and sensory functions, sexual function changes after spinal cord injury and is considered one of the most common problems, ranging from a decrease in sexual desire to disturbances of erection, orgasm and ejaculation.

Objective: To assess the impact of the complexity of traumatic spinal cord injury in male sexual function.

DETAILED DESCRIPTION:
Methods: Observational study (CEAC 41221414.5.0000.5208) conducted with 45 men, mean age 34 (CI 31.5 to 37.1), with spinal cord injury and active sex life. Sexual function was assessed by the International Index of Erectile Function (IIEF) and level and degree of injury were determined following the guidelines of the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury. Data were collected after at least six months of injury in referral hospitals. Descriptive statistics and bivariate analysis were applied to observe the association between sexual function and complexity of the lesion, with a 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* men
* aged between 18 and 60 years
* clinical diagnosis of traumatic spinal cord injury
* injury time equal to or greater than six months
* heterosexual
* sexually active.

Exclusion Criteria:

* patients with erectile dysfunction attributed to endocrine or metabolic disease order
* those who underwent surgery as radical prostatectomy or penile implant
* cognitive impairment.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Observational study, conducted between March 2015 and ending in January 2016, with males, aged between 18 and 60 years; clinical diagnosis of traumatic spinal cord injury, injury time equal to or greater than six months, heterosexual and sexually active.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sexual function | one day
  Sexual function assessed by the International Index of Erectile Function (IIEF)

SECONDARY OUTCOMES:
Degree of neurological lesion | one day
  Degree of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Level of neurological lesion | one day
  Level of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury

CONTACTS AND LOCATIONS:
Overall Officials: Josepha KO Ferro, master, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Josepha Karinne de Oliveira Ferro, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No